CLINICAL TRIAL: NCT03919331
Title: Impact of Current Volume Under High-rate Nasal Oxygen Therapy During Acute Hypoxemic Respiratory Failure de Novo
Acronym: IVOXY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP180138
Record Dates: First submitted 2019-03-26; First posted 2019-04-18 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-03

CONDITIONS: Acute Hypoxemic Respiratory Failure
Keywords: High flow nasal canula / P-SILI/ AHRF / EIT
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Tidal volume (TV) during high flow nasal canula (HFNC) will be measured using chest Electrical Impedance Tomography (EIT). To calibrate EIT data, i.e. to be able to convert changes in thoracic impedance into TV, thoracic impedance signal, flow and volume will be collected during a 4 cmH2O continuous positive airway pressure (CPAP) test, using a pneumotachograph inserted on the ventilator circuit between the mask and the Y-piece. Such a level of CPAP is supposed to reproduce the majority of the physiological effects of HFNC. The quantification of respiratory distress index will be recorded by respiratory inductance plethysmography (RIP), obtained using two elastic bands equipped with a sensor sensitive to their stretching, one positioned at the level of the thorax, the other at the level of the abdomen. The stretching changes of the two bands during the respiratory cycle allow evaluating their possible asynchronism by calculating the phase angle.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Every adult patient admitted to the medical intensive care unit for de novo acute hypoxemic respiratory failure, and placed under hign flow nasal canula (HFNC). Inclusion and exclusion criterion are listed elsewhere.
  Interventions: Diagnostic Test: Assessment of tidal volume using Electrical Impedance Tomography (EIT) during high flow nasal canula(HFNC)

INTERVENTIONS:
Diagnostic Test: Assessment of tidal volume using Electrical Impedance Tomography (EIT) during high flow nasal canula(HFNC) — After information and consent, patients under HFNC for de novo acute hypoxemic respiratory failure will undergo a ten minutes 4cmH2O continuous positive airway pressure(CPAP) test while monitored with 1)chest Electrical Impedance Tomography (EIT) 2) a pneumotachograph inserted on the ventilator circuit between the mask and the Y-piece and connected to a differential pressure sensor, and 3) respiratory inductance plethysmography (RIP). Airway flow signal will be acquired using an analog/digital converter and stored for further analysis with acknowledge software. This will allow converting EIT data into tidal volume (TV), and estimating TV under HFNC. RIP signals will allow evaluating asynchronism between chest and abdomen by calculating the phase angle, thus quantifying respiratory distress. Patients monitored with an arterial catheter, arterial blood gas measurements will be done during CPAP and HFNC. These measures will be collected the first day of HFNC, and everyday up to three days

SUMMARY:
De novo acute hypoxemic respiratory failure (AHRF) is associated with high overall mortality, which increases significantly with the use of orotracheal intubation. High flow nasal canula (HFNC) has turned to be the first line non-invasive oxygenation strategy aiming to avoid intubation. One of the main factors worsening lung injury and increasing mortality in invasively ventilated patients is a too high tidal volume (TV) delivered by the ventilator. Consistent data suggest that such an aggravation of respiratory lesions may occur during spontaneous ventilation if TV is too large. This phenomenon is called Patient self-inflicted lung injury (P-SILI). The effect of TV on the outcome of patients with de novo AHRF under HFNC has never been evaluated since TV is not easily accessible in patients under HFNC. Investigators hypothesized that a large TV during HFNC has an impact on the outcome. TV will be measured using chest Electrical Impedance Tomography (EIT). To calibrate the EIT data, i.e. to be able to convert changes in thoracic impedance into TV, thoracic impedance signal, flow and volume will be collected during a 4 cmH2O continuous positive airway pressure (CPAP) test, using a pneumotachograph inserted on the ventilator circuit between the mask and the Y-piece. Such a level of CPAP is supposed to reproduce the majority of the physiological effects of HFNC. Thus, EIT signal can be used to calculate TV during HFNC since it remains reliable even when the positive expiratory pressure changes.

A secondary objective is to quantify a respiratory distress index. This quantification will be recorded by respiratory inductance plethysmography (RIP), obtained using two elastic bands equipped with a sensor sensitive to their stretching, one positioned at the level of the thorax, the other at the level of the abdomen. The stretching changes of the two bands during the respiratory cycle allow evaluating their possible asynchronism by calculating the phase angle Investigators want to be able to evaluate up to 6 predictors of HFNC failure in this research with an effect size of 0.15, α risk of 0.05, and a power of 0.8. A number of 55 participants is required. Investigators plan to include 60 patients due to potential withdrawal of consent and/or unusable data.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* HFNC initiated as part of the care
* Respiratory rate > 25 / minute
* PaO2/FiO2 ratio < 300 mm Hg
* PaCO2 < 45 mm Hg
* Affiliated with a social security system
* Informed consent signed by the patient, trusted person or family member if the patient is unable to consent

Exclusion Criteria:

* Acute cardiogenic pulmonary edema
* Underlying chronic respiratory disease
* Asthma exacerbation
* Chronic obstructive pulmonary disease Exacerbation
* Hemodynamic instability, defined as systolic arterial blood pressure < 90 mm Hg or mean arterial blood pressure < 65 mm Hg or the use of vasopressors
* Glasgow Coma Score <= 12
* Contraindication to CPAP (maxillofacial surgery, facial trauma)
* Refusal of the patient to perform the CPAP test
* Need for emergency intubation according to the clinician in charge of the patient
* Patient protected by law
* Pregnancy or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2021-06-03 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Failure of high flow nasal canula (HFNC) at day 28 | Day 28
  Failure of HFNC is defined as death or need for invasive mechanical ventilation

SECONDARY OUTCOMES:
Tidal volume under high flow nasal canula (HFNC) | Day 0, Day 1 and Day 2
  Tidal volume will be measured using chest Electrical Impedance Tomography (EIT)
Phase angle computed by respiratory inductance plethysmography (RIP) | Day 0, Day 1 and Day 2
  Phase angle will be measured by respiratory inductance plethysmography
Respiratory rate | Day 0, Day 1 and Day 2
  respiratory rate will be measured at each evaluation
pH under high flow nasal canula (HFNC) | Day 0, Day 1 and Day 2
  pH will be measured via Blood gases
PaO2 under high flow nasal canula (HFNC) | Day 0, Day 1 and Day 2
  PaO2 will be measured via Blood gases
PaCO2 under high flow nasal canula (HFNC) | Day 0, Day 1 and Day 2
  PaCO2 will be measured via Blood gases
SaO2 under high flow nasal canula (HFNC) | Day 0, Day 1 and Day 2
  SaO2 will be measured via Blood gases
Regional tidal volume. | Day 0, Day 1 and Day 2
  computed by Electrical Impedance Tomography
Mortality | Day 28, Day90
  Mortality at Day 28, Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume CARTEAUX, Doctor, Principal Investigator — Assistance Publique Hôpitaux de Paris - CHU Henri Mondor - Créteil
Locations (1):
- Assistance Publique Hôpitaux de Paris - CHU Henri Mondor - Créteil, Créteil, France

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWN BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION

REFERENCES:
- [Background] Antonelli M, Conti G, Rocco M, Bufi M, De Blasi RA, Vivino G, Gasparetto A, Meduri GU. A comparison of noninvasive positive-pressure ventilation and conventional mechanical ventilation in patients with acute respiratory failure. N Engl J Med. 1998 Aug 13;339(7):429-35. doi: 10.1056/NEJM199808133390703. PMID 9700176
- [Background] Antonelli M, Conti G, Moro ML, Esquinas A, Gonzalez-Diaz G, Confalonieri M, Pelaia P, Principi T, Gregoretti C, Beltrame F, Pennisi MA, Arcangeli A, Proietti R, Passariello M, Meduri GU. Predictors of failure of noninvasive positive pressure ventilation in patients with acute hypoxemic respiratory failure: a multi-center study. Intensive Care Med. 2001 Nov;27(11):1718-28. doi: 10.1007/s00134-001-1114-4. Epub 2001 Oct 16. PMID 11810114
- [Background] Confalonieri M, Potena A, Carbone G, Porta RD, Tolley EA, Umberto Meduri G. Acute respiratory failure in patients with severe community-acquired pneumonia. A prospective randomized evaluation of noninvasive ventilation. Am J Respir Crit Care Med. 1999 Nov;160(5 Pt 1):1585-91. doi: 10.1164/ajrccm.160.5.9903015. PMID 10556125
- [Background] Frat JP, Thille AW, Mercat A, Girault C, Ragot S, Perbet S, Prat G, Boulain T, Morawiec E, Cottereau A, Devaquet J, Nseir S, Razazi K, Mira JP, Argaud L, Chakarian JC, Ricard JD, Wittebole X, Chevalier S, Herbland A, Fartoukh M, Constantin JM, Tonnelier JM, Pierrot M, Mathonnet A, Beduneau G, Deletage-Metreau C, Richard JC, Brochard L, Robert R; FLORALI Study Group; REVA Network. High-flow oxygen through nasal cannula in acute hypoxemic respiratory failure. N Engl J Med. 2015 Jun 4;372(23):2185-96. doi: 10.1056/NEJMoa1503326. Epub 2015 May 17. PMID 25981908
- [Background] Carteaux G, Millan-Guilarte T, De Prost N, Razazi K, Abid S, Thille AW, Schortgen F, Brochard L, Brun-Buisson C, Mekontso Dessap A. Failure of Noninvasive Ventilation for De Novo Acute Hypoxemic Respiratory Failure: Role of Tidal Volume. Crit Care Med. 2016 Feb;44(2):282-90. doi: 10.1097/CCM.0000000000001379. PMID 26584191
- [Background] Frat JP, Ragot S, Coudroy R, Constantin JM, Girault C, Prat G, Boulain T, Demoule A, Ricard JD, Razazi K, Lascarrou JB, Devaquet J, Mira JP, Argaud L, Chakarian JC, Fartoukh M, Nseir S, Mercat A, Brochard L, Robert R, Thille AW; REVA network. Predictors of Intubation in Patients With Acute Hypoxemic Respiratory Failure Treated With a Noninvasive Oxygenation Strategy. Crit Care Med. 2018 Feb;46(2):208-215. doi: 10.1097/CCM.0000000000002818. PMID 29099420
- [Background] Brochard L, Slutsky A, Pesenti A. Mechanical Ventilation to Minimize Progression of Lung Injury in Acute Respiratory Failure. Am J Respir Crit Care Med. 2017 Feb 15;195(4):438-442. doi: 10.1164/rccm.201605-1081CP. PMID 27626833
- [Background] Chanques G, Riboulet F, Molinari N, Carr J, Jung B, Prades A, Galia F, Futier E, Constantin JM, Jaber S. Comparison of three high flow oxygen therapy delivery devices: a clinical physiological cross-over study. Minerva Anestesiol. 2013 Dec;79(12):1344-55. Epub 2013 Jul 15. PMID 23857440
- [Background] Mauri T, Eronia N, Turrini C, Battistini M, Grasselli G, Rona R, Volta CA, Bellani G, Pesenti A. Bedside assessment of the effects of positive end-expiratory pressure on lung inflation and recruitment by the helium dilution technique and electrical impedance tomography. Intensive Care Med. 2016 Oct;42(10):1576-1587. doi: 10.1007/s00134-016-4467-4. Epub 2016 Aug 12. PMID 27518321
- [Background] Hammer J, Newth CJ. Assessment of thoraco-abdominal asynchrony. Paediatr Respir Rev. 2009 Jun;10(2):75-80. doi: 10.1016/j.prrv.2009.02.004. Epub 2009 Apr 9. PMID 19410206
- [Derived] Tuffet S, Boujelben MA, Haudebourg AF, Maraffi T, Perier F, Labedade P, Moncomble E, Gendreau S, Lacheny M, Vivier E, Mekontso-Dessap A, Carteaux G. High flow nasal cannula and low level continuous positive airway pressure have different physiological effects during de novo acute hypoxemic respiratory failure. Ann Intensive Care. 2024 Nov 23;14(1):171. doi: 10.1186/s13613-024-01408-w. PMID 39578265